CLINICAL TRIAL: NCT06213194
Title: Investigating The Effects of Executive Functions and Social Cognition on the Relationship Between Autistic Traits and Mental Health
Brief Title: The Effects of Executive Functions and Social Cognition on Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Haldun University (Other)
Responsible Party: Principal Investigator, Dilruba Sönmez, Clinical Psychologist, Ibn Haldun University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/07-03
Record Dates: First submitted 2023-12-14; First posted 2024-01-19 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Autism or Autistic Traits; Mental Health Disorder; Executive Dysfunction; Social Cognition
Keywords: Autism; Executive Functions; Online Training; Social Cognition; Mental Health
MeSH Terms: conditions — Autistic Disorder; Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: All participants would be assigned randomly to the experimental group and control group (wait-list condition) to see whether the combined training program is effective for the general population.
Who Masked: Participant
Masking Description: To reduce biases, a single-blind procedure will be applied. It will be provided basic information about topics including social-cognitive skills and mental health but no detailed description of training will be given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): It combines social cognitive and executive functions skills and it will be present on the designed website and they will participate in the intervention online. After participants are assigned the experimental group the 6-week training program will start and they cannot access the next week before completing the previous week. Each week's will last about 75 minutes. The training includes social cognitive skills including cognitive and affective empathy and executive functions.
  Interventions: Other: MindZone
- Control Group (No Intervention): This group will not take the training until the follow-up test. After the study will be done, the training program will be offered to the control group as well.

INTERVENTIONS:
Other: MindZone — The name of the online training will be MindZone. It consists of combined game-based social cognitive and executive functions skills, and it will be presented on the training website. There is no consensus about the length of time for the training in the literature, so the average time for the training process will be used. This means that the training will last 6 weeks, 7.5 hours in total. To satisfy the training requirement, 1.15 hours (75 mins) of play will be expected from participants each week. Before each game, a brief introduction about the game will be presented and participants will get feedback about their progress. Each participant will conduct the tasks in a different random order. After 6 weeks, a post-test will be completed, and follow-up scores will be obtained after a month. All tasks were designed according to the five intervention areas: working memory, cognitive flexibility, inhibition, cognitive empathy and affective empathy based on the literature.
  Arms: Experimental Group

SUMMARY:
The objective of this study is to analyze the effects of executive functions (EFs) and social-cognitive abilities on the associations between autistic traits and mental health indicators (depression, anxiety, and stress). Moreover, the study will produce online training modules for executive functions and social cognition, aimed at reducing the likelihood of adverse mental health outcomes in individuals with and without elevated autistic traits.

Therefore, four main hypotheses will be addressed:

1. Revealing the mediating role of executive functions (cognitive flexibility, inhibitory control, and working memory) will help predict the association between autistic traits and mental health symptoms (anxiety, depression, and stress).
2. Revealing the mediating role of social cognitive skills (cognitive empathy and affective empathy) will help predict the association between autistic traits and mental health symptoms (anxiety, depression, and stress).
3. Online training in executive functions and social cognitive skills will help develop executive functions (working memory, inhibitory control, and cognitive flexibility) and social cognitive skills (cognitive empathy and affective empathy) in the current sample.
4. Online training in executive functions and social cognitive skills will promote mental health by reducing distress, depression, and anxiety symptoms in the current sample.

Participants will be between the ages of 18-35 because previous findings indicate that the age of onset of various mental health problems is between the ages of 17 and 35. Participants will be randomly assigned to the experimental and control groups. Using a longitudinal design including pre-test, post-test, and follow-up conditions to test the effectiveness of combined EFs and social cognition online training for mental health symptoms.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) refers to a neurodevelopmental condition that is associated with impairments in social and cognitive functions, repetitive behaviors, and restricted interests, while autistic traits refer to a subclinical level of ASD and its symptoms distributed in the general population. Previous studies have identified people with elevated autistic traits who show susceptibility to other mental health conditions such as anxiety disorders, mood disorders, borderline personality disorder, internet addiction, conduct disorder, substance abuse, and suicidal risk in the general population. Although there is no identifiable explanation of susceptibility to other mental health conditions, the presence of social and cognitive impairments including problems in executive functions and social cognitive skills might be contributing factors.

Previous research indicated that social cognitive skills such as cognitive and affective empathy and executive functions including working memory, inhibitory control and cognitive flexibility play important roles in physical and mental health, quality of life, social competence, school and job success, marital harmony, and public safety. Nevertheless, although autistic traits increase susceptibility to other mental health conditions, no study so far has focused on examining the relationships among autistic traits, executive functions, and social cognitive skills to design intervention and prevention programs for mental health conditions and quality of life in both general and clinical populations.

The primary purpose of the research is to investigate the effects of executive functions and social cognitive skills on the relationship between autistic traits and mental health symptoms that would be significant for designing intervention and prevention programs. The second purpose of the research is to design online executive functions and social cognitive training that might help to reduce vulnerability to negative effects on mental health symptoms in the general population regarding elevated autistic traits.

Using a longitudinal design including pre-test, post-test, and follow-up conditions to test the effectiveness of combined executive functions (EFs) and social cognition online training via computers, tablets, or smartphones for mental health symptoms (depression, anxiety, and stress). This study's independent variables are executive functions (cognitive flexibility, inhibition, and working memory) and social cognition (cognitive empathy and affective empathy). Dependent variables are mental health scores (depression, anxiety, and stress symptoms). Participants will be between the ages of 18 and 35 because previous findings indicate that the age of onset of various mental health problems is between the ages of 17 and 35. Participants will be randomly assigned to the experimental and control groups. Online-based training will consist of combined executive functions and social cognitive (i.e., cognitive empathy and affective empathy) tasks. The length of the training each week will be 75 minutes based on the previous studies. Three within conditions will be present: pre-test, post-test, and follow-up. The primary outcomes of the study are mental health symptoms (anxiety, depression, stress), EFs (working memory, cognitive flexibility, and inhibition), and social cognition (cognitive and affective empathy).

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 or above
2. Fluent in writing and speaking in Turkish
3. No record of any psychiatric disorders
4. No record of neurological conditions

Exclusion Criteria:

1. under age 18
2. Have any record of psychiatric
3. Have any neurological conditions

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dilruba Sönmez, MA, Principal Investigator — Ibn Haldun University
Locations (1):
- Dilruba Sönmez, Istanbul, Basaksehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
To ensure the ethical rights of the participants, the data will be available only for current research unless the participants give permission.

REFERENCES:
- [Background] Sonmez D, Jordan TR. Investigating associations between cognitive empathy, affective empathy and anxiety in adolescents with autism spectrum disorder. Int J Dev Disabil. 2023 Jan 9;70(5):957-965. doi: 10.1080/20473869.2022.2163605. eCollection 2024. PMID 39131758
- [Result] Albantakis L, Brandi ML, Zillekens IC, Henco L, Weindel L, Thaler H, Schliephake L, Timmermans B, Schilbach L. Alexithymic and autistic traits: Relevance for comorbid depression and social phobia in adults with and without autism spectrum disorder. Autism. 2020 Nov;24(8):2046-2056. doi: 10.1177/1362361320936024. Epub 2020 Jul 14. PMID 32662285
- [Result] Baron-Cohen S. The extreme male brain theory of autism. Trends Cogn Sci. 2002 Jun 1;6(6):248-254. doi: 10.1016/s1364-6613(02)01904-6. PMID 12039606
- [Result] Craig F, Margari F, Legrottaglie AR, Palumbi R, de Giambattista C, Margari L. A review of executive function deficits in autism spectrum disorder and attention-deficit/hyperactivity disorder. Neuropsychiatr Dis Treat. 2016 May 12;12:1191-202. doi: 10.2147/NDT.S104620. eCollection 2016. PMID 27274255
- [Result] Dell'Osso L, Carpita B, Muti D, Morelli V, Salarpi G, Salerni A, Scotto J, Massimetti G, Gesi C, Ballerio M, Signorelli MS, Luciano M, Politi P, Aguglia E, Carmassi C, Maj M. Mood symptoms and suicidality across the autism spectrum. Compr Psychiatry. 2019 May;91:34-38. doi: 10.1016/j.comppsych.2019.03.004. Epub 2019 Apr 3. PMID 31003723
- [Result] de Vries M, Prins PJ, Schmand BA, Geurts HM. Working memory and cognitive flexibility-training for children with an autism spectrum disorder: a randomized controlled trial. J Child Psychol Psychiatry. 2015 May;56(5):566-76. doi: 10.1111/jcpp.12324. Epub 2014 Sep 26. PMID 25256627
- [Result] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Result] Fietz J, Valencia N, Silani G. Alexithymia and autistic traits as possible predictors for traits related to depression, anxiety, and stress: A multivariate statistical approach. J Eval Clin Pract. 2018 Aug;24(4):901-908. doi: 10.1111/jep.12961. Epub 2018 Jun 8. PMID 29882629
- [Result] Gambin M, Sharp C. Relations between empathy and anxiety dimensions in inpatient adolescents. Anxiety Stress Coping. 2018 Jul;31(4):447-458. doi: 10.1080/10615806.2018.1475868. Epub 2018 May 17. PMID 29772912
- [Result] Gardiner E, Iarocci G. Everyday executive function predicts adaptive and internalizing behavior among children with and without autism spectrum disorder. Autism Res. 2018 Feb;11(2):284-295. doi: 10.1002/aur.1877. Epub 2017 Sep 27. PMID 28960841
- [Result] Gokcen E, Frederickson N, Petrides KV. Theory of Mind and Executive Control Deficits in Typically Developing Adults and Adolescents with High Levels of Autism Traits. J Autism Dev Disord. 2016 Jun;46(6):2072-2087. doi: 10.1007/s10803-016-2735-3. PMID 26886468
- [Result] Lundstrom S, Chang Z, Kerekes N, Gumpert CH, Rastam M, Gillberg C, Lichtenstein P, Anckarsater H. Autistic-like traits and their association with mental health problems in two nationwide twin cohorts of children and adults. Psychol Med. 2011 Nov;41(11):2423-33. doi: 10.1017/S0033291711000377. Epub 2011 Mar 22. PMID 21426604
- [Result] Mason D, Happe F. The role of alexithymia and autistic traits in predicting quality of life in an online sample. Res Autism Spectr Disord. 2022 Feb;90:None. doi: 10.1016/j.rasd.2021.101887. PMID 35116075
- [Result] Nahum M, Lee H, Fisher M, Green MF, Hooker CI, Ventura J, Jordan JT, Rose A, Kim SJ, Haut KM, Merzenich MM, Vinogradov S. Online Social Cognition Training in Schizophrenia: A Double-Blind, Randomized, Controlled Multi-Site Clinical Trial. Schizophr Bull. 2021 Jan 23;47(1):108-117. doi: 10.1093/schbul/sbaa085. PMID 32614046
- [Result] Sandgreen H, Frederiksen LH, Bilenberg N. Digital Interventions for Autism Spectrum Disorder: A Meta-analysis. J Autism Dev Disord. 2021 Sep;51(9):3138-3152. doi: 10.1007/s10803-020-04778-9. Epub 2020 Nov 10. PMID 33170393
- [Result] Sari BA, Koster EH, Pourtois G, Derakshan N. Training working memory to improve attentional control in anxiety: A proof-of-principle study using behavioral and electrophysiological measures. Biol Psychol. 2016 Dec;121(Pt B):203-212. doi: 10.1016/j.biopsycho.2015.09.008. Epub 2015 Sep 25. PMID 26407521
- [Result] Zelazo PD. Executive Function and Psychopathology: A Neurodevelopmental Perspective. Annu Rev Clin Psychol. 2020 May 7;16:431-454. doi: 10.1146/annurev-clinpsy-072319-024242. Epub 2020 Feb 19. PMID 32075434
- [Result] Allemand M, Steiger AE, Fend HA. Empathy development in adolescence predicts social competencies in adulthood. J Pers. 2015 Apr;83(2):229-41. doi: 10.1111/jopy.12098. Epub 2014 May 4. PMID 24684661
- [Result] Eussen ML, Van Gool AR, Verheij F, De Nijs PF, Verhulst FC, Greaves-Lord K. The association of quality of social relations, symptom severity and intelligence with anxiety in children with autism spectrum disorders. Autism. 2013 Nov;17(6):723-35. doi: 10.1177/1362361312453882. Epub 2012 Aug 23. PMID 22917843
- [Result] Solmi M, Radua J, Olivola M, Croce E, Soardo L, Salazar de Pablo G, Il Shin J, Kirkbride JB, Jones P, Kim JH, Kim JY, Carvalho AF, Seeman MV, Correll CU, Fusar-Poli P. Age at onset of mental disorders worldwide: large-scale meta-analysis of 192 epidemiological studies. Mol Psychiatry. 2022 Jan;27(1):281-295. doi: 10.1038/s41380-021-01161-7. Epub 2021 Jun 2. PMID 34079068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Online data collection were used.
Pre-assignment Details: Participants are under the age of 18, and who have any record of psychiatric or physical conditions excluded from the study.
Groups:
- Experimental Group: It combines social cognitive and executive functions skills and it will be present on the designed website and they will participate in the intervention online. After participants are assigned the experimental group the 6-week training program will start and they cannot access the next week before completing the previous week. Each week's will last about 75 minutes. The training includes social cognitive skills including cognitive and affective empathy and executive functions.
  MindZone: The name of the online training will be MindZone. It consists of combined game-based social cognitive and executive functions skills, and it will be presented on the training website. There is no consensus about the length of time for the training in the literature, so the average time for the training process will be used. This means that the training will last 6 weeks, 5 hours in total. To satisfy the training requirement, 50 mins for each week of play will be expected from participants each week. Before each game, a brief introduction about the game will be presented and participants will get feedback about their progress. Each participant will conduct the tasks in a different random order. After 6 weeks, a post-test will be completed, and follow-up scores will be obtained after a month. All tasks were designed according to the five intervention areas: working memory, cognitive flexibility, inhibition, cognitive empathy and affective empathy based on the literature.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 89 | 89
Completed | 31 | 34
Not Completed | 58 | 55

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 89 | 89 | 178
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 89 | 178
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: We included participants who completed the post-test condition.
  years
    number analyzed (Participants) | 31 | 34 | 65
    (all) | 27.58 (5.95) | 27.24 (6.13) | 27.41 (6.02)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We included the participants who completed the post-test condition.
  Participants
    number analyzed (Participants) | 31 | 34 | 65
    Female | 28 | 29 | 57
    Male | 3 | 5 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 89 | 89 | 178

OUTCOME MEASURES:

1. Primary Outcome: Depression_1
Description: Depression Anxiety Stress Scale 21 will be used to measure depression outcome. Higher scores mean higher depressive symptoms. The minimum and maximum scores are 0-21, respectively.
Time Frame: Pre-test (baseline), Post-test (immediately after the intervention)
Population: Experimental and control groups
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Group: Pretest Mean (SD) :9.87(3.72) Posttest Mean (SD): 7.65 (2.57)
- Control Group: depression subscale of DASS-21
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 34
score on a scale
  Pretest | 9.87 (3.72) | 10.24 (4.02)
  Posttest | 7.65 (2.57) | 9.15 (4.13)

2. Primary Outcome: Anxiety
Description: Depression Anxiety Stress Scale - 21 will be used to measure anxiety outcome. Higher scores mean higher anxiety symptoms. The minimum and maximum scores are 0-21, respectively.
Time Frame: Pre-test (baseline), Post-test (immediately after the intervention)
Population: experimental and control groups
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Group: Anxiety subscale, pretest and posttest condition. Pretest:9.42 (3.70) Posttest:6.74 (2.94)
- Control Group: anxiety subscale from DASS-21
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 34
score on a scale
  Pretest | 9.42 (3.70) | 9.44 (3.94)
  Posttest | 6.74 (2.94) | 8.03 (4.20)

3. Primary Outcome: Stress
Description: Depression Anxiety Stress Scale - 21 will be used to measure stress outcome. Higher scores indicate higher stress. The minimum and maximum scores are 0-21, respectively.
Time Frame: Pre-test (baseline), Post-test (immediately after the intervention)
Population: experimental group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Group: Stress subscale
- Control Group: stress subscale of DASS-21
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 34
score on a scale
  Pretest | 7.61 (3.98) | 6.32 (3.98)
  Posttest | 5.58 (3.56) | 7.79 (4.05)

4. Primary Outcome: Cognitive Flexibility - Errors Rate
Description: Cognitive flexibility - Errors Rate will be measured by the Wisconsin Card Sorting Task. Higher errors indicate lower scores on cognitive flexibility. During the task, 400 cards in two blocks are displayed on the screen and the sorting rule changes after every 10 cards. Maximum score is 400 and minimum score is 0.
Time Frame: Pre-test (baseline), Post-test (immediately after the intervention)
Population: experimental group vs. control group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Group: Cognitive flexbility - errors
- Control Group: Control group error scores
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 34
score on a scale
  Pretest | 21 (10) | 22 (4)
  Posttest | 40 (20) | 37 (15)

5. Primary Outcome: Working Memory - Errors Rate
Description: Working memory - Errors Rate will be measured by the N-back task. Higher errors indicate lower working memory scores. Maximum score is 400, minimum score is 0
Time Frame: Pre-test (baseline), Post-test (immediately after the intervention)
Population: experimental group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Group: Errors rate
- Control Group: Control group errors scores
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 34
score on a scale
  Pretest | 20.65 (9.19) | 15.09 (11.94)
  Posttest | 13.13 (8.59) | 10.50 (7.55)

6. Primary Outcome: Inhibition - Errors Rate
Description: Inhibition - Errors Rate will be measured by Go/No Go task. Higher scores indicate lower inhibition. There are 12 blocks of 50 trials each. Commission errors (i.e., incorrectly responding to no-go trials) were measured. Maximum score is 600. Minimum score is 0.
Time Frame: Pre-test (baseline), Post-test (immediately after the intervention)
Population: experimental group vs. control group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Group: Inhibitory Control - Errors rate
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 34
score on a scale
  Pretest | 5.48 (6.59) | 3.24 (5.18)
  Posttest | 4.48 (3.37) | 3.85 (3.21)

7. Secondary Outcome: Cognitive Empathy
Description: The Eyes Test were used to measure cognitive empathy. Higher scores indicate higher cognitive empathy scores. Maximum score is 36, minimum score is 0.
Time Frame: pretest and posttest conditions
Population: experimental and control groups
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Group; Control Group: accuracy
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 34
score on a scale
  Pretest | 24.45 (3.88) | 25.65 (3.27)
  Posttest | 25.39 (4.29) | 26.59 (3.44)

8. Secondary Outcome: Self-Assessment Manikin for Affective Empathy
Description: Self Assessment Manikin was used to measure affective empathy. Valence scores for each emotion were obtained by summing responses for all images. The maximum score is 270, and the minimum score is 30. Higher scores indicate better affective empathy.
Time Frame: pretest and posttest conditions
Population: experimental and control groups
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Group; Control Group: summing the scores for affective empathy performance task
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 34
score on a scale
  Pretest | 130.16 (20.43) | 119.35 (16.88)
  Posttest | 126.16 (12.90) | 117.38 (16.61)

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed.
Description: Adverse Events were not monitored/assessed.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT06213194/Prot_SAP_000.pdf